CLINICAL TRIAL: NCT01542463
Title: Levemir®: the Physiological Basal Insulin. Documentation of Safety Aspects, Glycaemic Control and Weight
Brief Title: Evaluation of the Use of Levemir® in Insufficiently Controlled Patients With Type 1 or Type 2 Diabetes
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: NN304-1893
Record Dates: First submitted 2012-02-24; First posted 2012-03-02 (Estimated); Last update posted 2016-03-03 (Estimated); Status verified 2016-03

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2 | interventions — Insulin Detemir

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- IDet users
  Interventions: Drug: insulin detemir

INTERVENTIONS:
Drug: insulin detemir — Prescribed at the discretion of the physician

SUMMARY:
This study conducted in Europe. The aim of this study is to evaluated the use of insulin detemir (Levemir®) in insufficiently controlled patients with type 1 or type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Patients with insufficiently controlled type 1 or type 2 diabetes mellitus under their previous therapy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with insufficiently controlled type 1 or type 2 diabetes mellitus under their previous therapy
Sampling Method: Non-Probability Sample
Enrollment: 4464 (Actual)
Dates: Start 2004-09; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
HbA1c (glycaemic haemoglobin)
Fasting plasma glucose (FBG)

SECONDARY OUTCOMES:
Body weight change
Adverse drug reactions (ADR)
Serious adverse drug reactions (SADR)
Hypoglycaemic episodes

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Mainz, Germany

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com